CLINICAL TRIAL: NCT00696826
Title: An Open-Label, Single Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of MK0431
Brief Title: A Study of MK0431 in Patients WIth Hepatic Insufficiency (0431-017)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-017; MK0431-017; 2008_530
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Liver Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Sitagliptin Phosphate

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin phosphate 100 mg MK0431 (2 x 50 mg tablets) taken orally after overnight fast; Duration of Treatment: 5 Weeks
  Other Names: MK0431

SUMMARY:
A study to compare the plasma concentrations of MK0431 at different times in patients with hepatic insufficiency vs healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* If female, non pregnant, BMI less than 40 kg/m2
* Patient has chronic, stable hepatic insufficiency

Exclusion Criteria:

* Patient unwilling to refrain from alcohol and grapefruit juice prior to and shortly after study drug administration
* Patient has diabetes, had a heart attack or stroke, or uncontrolled congestive heart failure during the past 6 months
* Patient has a history of drug or alcohol abuse
* Patient smokes > 10 cigarettes per day
* Patient consumes more that 6 cups of caffeinated beverages per day
* Patient has had surgery, donated blood or participated in another clinical trial within the past 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
the plasma and urine pharmacokinetic parameters of MK0431 | measured at predose, 0.5, 1,1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 18, 24, 32, 48, 72 and 96 hours post dose

SECONDARY OUTCOMES:
Side effects, physical exam, lab safety data, urging drug screen, ECG and vital signs | throughout study and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Migoya EM, Stevens CH, Bergman AJ, Luo WL, Lasseter KC, Dilzer SC, Davies MJ, Wagner JA, Herman GA. Effect of moderate hepatic insufficiency on the pharmacokinetics of sitagliptin. Can J Clin Pharmacol. 2009 Winter;16(1):e165-70. Epub 2009 Feb 16. PMID 19221403